CLINICAL TRIAL: NCT06352411
Title: Pharmacokinetics, Safety, and Tolerability of BI 456906 Following Subcutaneous Injection in Male and Female Participants With Mild, Moderate and Severe Renal Impairment in Comparison to Participants With Normal Renal Function (Mono-centric, Open-label Study With Parallel Matched-pair Design)
Brief Title: A Study to Test How BI 456906 is Taken up in the Blood of People With and Without Kidney Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0009; 2023-508557-13-00 (Registry Identifier: CTIS); U1111-1298-3135 (Registry Identifier: WHO registry)
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — BI 456906

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: Participants with normal renal function (Experimental)
  Interventions: Drug: BI 456906
- Group 2: Participants with mild renal impairment (Experimental)
  Interventions: Drug: BI 456906
- Group 3: Participants with moderate renal impairment (Experimental)
  Interventions: Drug: BI 456906
- Group 4: Participants with severe renal impairment (Experimental)
  Interventions: Drug: BI 456906

INTERVENTIONS:
Drug: BI 456906 — Solution for injection
  Other Names: survodutide

SUMMARY:
This study is open to adults aged between 18 and 80 years of age with a body mass index (BMI) of 20 to 40 kg/m2. People with or without kidney problems can take part in the study.

The purpose of this study is to find out how much of a medicine called BI 456906 gets into the blood of people with and without kidney problems. BI 456906 is being developed to treat people with obesity and liver problems. People living with these conditions often also have kidney problems. Therefore, it is important to find out whether kidney problems influence the amount of BI 456906 that gets into the blood.

Study participants receive a single dose of BI 456906 as an injection under the skin. Participants are divided into 4 groups based on how well their kidneys work: 1 group without kidney problems, and 3 groups with mild, moderate, and severe kidney problems. Each participant without kidney problems is matched with participants from the other groups based on factors such as age, gender, race, and body mass index (BMI) to ensure accurate comparisons.

Participants are in the study for about 2 months. They stay for 5 days and 4 nights at the study site and visit their doctors about 7 times. During these visits, the doctors collect information about participants' health. To assess the study endpoints, the doctors regularly take blood samples from the participants. The participants also answer questions about their well-being. The doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria applicable to all participants

Participants will only be included in the trial if they meet the following criteria:

* Male or female participants with age 18 to 80 years, inclusive at the screening visit.
* Body mass index (BMI) of 20.0-40.0 kg/m^2 (inclusive).
* Signed and dated written informed consent in accordance with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use -good clinical practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male participants are not required to use contraception. Further criteria apply.

Inclusion criteria applying only to participants with impaired renal function:

* Renal impairment based on assessment of estimated glomerular filtration rate (eGFR) at screening (severe renal impairment: 10.0-29.9 mL/min, moderate renal impairment: 30.0 - 59.9 mL/min (with at least 4 participants with a GFR between 30.0 and 45.0 mL/min), mild renal impairment: 60.0 - 89.9 mL/min)
* Chronic renal impairment > 12 months (documented renal impairment indicated by reduced eGFR for more than 12 months until screening)
* Absence of clinically significant abnormalities, as based on a complete medical history including a full physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests at screening, with the exception of findings that in the opinion of the investigator are consistent with the participant's renal impairment.
* Medication and/or treatment regimens must have been stable (i.e., no dose adjustments) for at least 4 weeks prior to the screening period and should be kept stable until study completion. Fluctuating treatment regimens may be considered for inclusion on a case-by-case basis if the underlying disease is under control in the opinion of the investigator and must be agreed to by both the investigator and the sponsor's medical monitor. Further criteria apply.

Exclusion criteria applying to all participants

* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Diseases of the central nervous system (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections Further criteria apply.

Exclusion criteria applying only to participants with renal impairment

* A marked prolongation of ECG interval from the start of the QRS complex (measured from the beginning of the Q wave to the end of the S wave) to the end of the T wave (QT)/QT interval corrected for heart rate, e.g. using the method of Fridericia (QTcF) or Bazett (QTcB)(QTc) interval (such as QTc intervals that are repeatedly greater than 480 milliseconds (ms) in males or repeatedly greater than 500 ms in females) or any other relevant ECG finding at screening
* Acute renal failure or active nephritis
* Nephrotic syndrome
* Impaired hepatic function, including relevant increases in liver enzymes indicating liver disease Further criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 456906 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to Day 29
Maximum measured concentration of BI 456906 in plasma (Cmax) | up to Day 29

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 456906 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to Day 29
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 36 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - CRS Clinical Research Services Mannheim GmbH, Mannheim

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com